CLINICAL TRIAL: NCT02957435
Title: Phase I, Open-label, Three Periods Study in Health Male and Female Subjects, Under Fasting Condition for Evaluation of Pharmacokinetics Profile of Single Dose of Eplerenone in Coated Tablets Formulation on Concentrations of 25mg, 50mg and 100mg, Produced by Biolab Sanus Farmacêutica Ltda
Brief Title: Pharmacokinetics Study of Eplerenone Coated Tablets
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Study has been cancelled and it has not been initiated.
Sponsor: Biolab Sanus Farmaceutica (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CAEP 56.005.16
Record Dates: First submitted 2016-11-03; First posted 2016-11-07 (Estimated); Last update posted 2018-06-06 (Actual); Status verified 2018-05

CONDITIONS: Pharmacokinetics; Healthy Subjects; Fasting
MeSH Terms: conditions — Fasting | interventions — Eplerenone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- eplerenone (Experimental): (Single arm) Sequence 1: one eplerenone coated tablet 25 mg in fasting (period 1), one eplerenone coated tablet 50 mg in fasting (period 2) and two eplerenone coated tablets 50 mg (100 mg of eplerenone) in fasting (period 3)
  Interventions: Drug: eplerenone

INTERVENTIONS:
Drug: eplerenone — (Single arm) Sequence 1: one eplerenone coated tablet 25 mg in fasting (period 1), one eplerenone coated tablet 50 mg in fasting (period 2) and two eplerenone coated tablets 50 mg (100 mg of eplerenone) in fasting (period 3)

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetics profile of the formulation of eplerenone coated tablets in the concentration of 25mg, 50mg and 100mg (2 coated tablets of 50mg) in male and female healthy subjects under fasting condition.

DETAILED DESCRIPTION:
This is a phase I study of eplerenone coated tablets of 25mg, 50mg and 100mg (2 coated tablets of 50mg) in fasting administration. Sample size is 12 subjects, male and female, aged between 18 and 50 years old.

This is an open-label, unicenter study with three periods, three treatments and one sequence. Each subject will receive the following treatments at the following periods:

* Period 1: one coated tablet of eplerenone 25mg in fasting
* Period 2: one coated tablet of eplerenone 50mg in fasting
* Period 3: two coated tablets of eplerenone 50mg (100mg of eplerenone) in fasting Formulations will be administered in a single dose, orally in each period. Trial subjects will be admitted in three different periods of 24 hours each, when investigational product will be administered and blood samples will be collected at pre-determined periods of time for pharmacokinetics evaluation.

Primary objective is to evaluate the pharmacokinetics of formulations of eplerenone coated tablets of 25mg, 50mg and 100mg (two coated tablets of 50mg) in healthy subjects under fasting condition. As a secondary objective, it will be also evaluated the safe and tolerability of coated tablets of eplerenone.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects, with age between 18 and 50 years old;
* Body mass index (BMI) between 18.5 and 30 kg/m2;
* Good health conditions or without significant diseases, at investigator discretion, according to the protocol and evaluation performed such as: clinical history, vital signs, physical examination, electrocardiogram (ECG) and laboratory exams;
* Ability to understand the nature and the objective of the trial, including risks and adverse effects.

Exclusion Criteria:

* Know hypersensitivity to the investigational product (eplerenone) or chemically related compounds;
* History or presence of chronic hepatic or gastrointestinal diseases, or other condition that may interfere with drug absorption, distribution, metabolism or excretion;
* Be in use of maintenance therapy with any drugs that interferes with the investigational product, except oral contraceptives;
* History of hepatic, kidney, lungs, gastrointestinal, epileptic, hematologic, psychiatric diseases, hypertension of any etiology, history of myocardial infarction, angina and/or heart failure or malignant neoplasias, in other words, any current disease, acute or chronic, in monitoring or treatment;
* Electrocardiographic findings that at investigator discretion are not recommended for study participation;
* History of any cardiac surgery, kidney surgery (exeresis or kidney anegesis), intestinal (partial or full ablation of esophagus, stomach, duodenum, jejunum, ileum, ascending colon, transverse colon, descending colon, sigmoid or rectum) and liver or pancreas surgery;
* Laboratory exams results out of the range considered normal in accordance with the reference ranges stipulated by the clinical laboratory, unless that are considered as not clinically significant by the investigator);
* Be a smoker;
* Ingestion of food that contains xanthine including more than five cups of coffee or tea per day;
* Vegan habits;
* History of abusive use of drugs and/or alcohol or excessive alcohol consumption;
* Have used regular medication in two weeks prior to start of treatment and the date of evaluation or have used any medication one week before, except contraceptives or in cases that, based on the half-life of the drug and/or active metabolites may be assumed the complete elimination;
* Have been hospitalized for any reason up to 8 weeks prior to start of the first period of trial treatment;
* Have received any treatment with any drug with known and well-established toxic potential to major organs inside of the 3 months prior to the study;
* Have participated from any experimental trial or have ingested any investigational drug within 12 months prior to the trial start;
* Be pregnant or in breastfeeding period or want to get pregnant during the study period;
* Have donated or have lost 450 mL or more of blood within 3 months prior to the trial or donation of more than 1500 mL of blood within 12 months prior to the trial;
* Have any condition, that prohibits the subject to participate in the trial, at the investigator's discretion;
* Have difficulty to swallow medicines and/or approximately 200 mL of water at the morning;
* Inability to keep awake or seated during one hour or necessary time at investigator discretion;
* Present a positive pregnancy test;
* Present breathalyzer test higher than zero;
* Present a positive result for a preliminary test of drugs.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2017-07 (Estimated); Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Maximum serum concentration (Cmax) | 24 hours
Area under the curve (ASCo-t) | 24 hours

SECONDARY OUTCOMES:
Time to reach Cmax (Tmax) | 24 hours
Half-life (t1/2) | 24 hours
Elimination constant rate (Kel) | 24 hours
Area under the curve (0-inf) | 24 hours
Number of adverse events | 30 days
Intensity of adverse events | 30 days
Causality of adverse events | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Pedro S Junior, MD, Principal Investigator — CAEP - Centro Avançado de Estudos e Pesquisa Ltda.
Locations (1):
- CAEP - Centro Avançado de Estudos e Pesquisas Ltda., Campinas, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No